CLINICAL TRIAL: NCT00883038
Title: Does a Low-Fat Vegetarian Diet Improve Insulin Resistance in Individuals With Type 2 Diabetes?
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Institute for Clinical and Experimental Medicine (Other Government)
Responsible Party: Dagmar Koveslygetyova, Institute for Clinical and Experimental Medicine
Allocation: Randomized | Model: Parallel | Purpose: Treatment
Other Study IDs: 785206
Record Dates: First submitted 2008-07-15; First posted 2009-04-17 (Estimated); Last update posted 2009-04-17 (Estimated); Status verified 2009-04

CONDITIONS: Insulin Resistance
Keywords: insulin resistance; vegetarian diet
MeSH Terms: conditions — Insulin Resistance

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Active Comparator (Active Comparator): Diabetic diet following the DNSG guidelines
  Interventions: Other: diabetic diet following the DNSG guidelines
- Experimental (Experimental): Low-fat vegetarian diet
  Interventions: Other: low-fat vegetarian diet

INTERVENTIONS:
Other: diabetic diet following the DNSG guidelines — The DNSG diet consists of 15-20% protein, ≤7% saturated fat, 60-70% carbohydrate and monounsaturated fats, cholesterol ≤200 mg/day, fiber content 20-30g/day.
  Arms: Active Comparator
Other: low-fat vegetarian diet — The low-fat vegetarian diet (~10% of energy from fat, 15% protein, and 75% carbohydrate, fiber content 40-50 g/day) consists of vegetables, fruits, grains, legumes and small amounts of nuts. Participants will be asked to avoid animal products and added fats and to favor low-glycemic index foods, such as beans and green vegetables.
  Arms: Experimental

SUMMARY:
The aim of the study is to evaluate the effect of experimental (vegetarian) diet compared to conventional diet with similar caloric restriction on insulin resistance, body weight and body composition in type 2 diabetic patients after 3 month diet program and additional 3 month diet program combined with intensive exercise.

Hypothesis: Greater improvement in insulin resistance, greater weight loss without compromising the body composition (subjects will lose fat preferentially to lean body mass) and differences in the fatty tissue metabolism will be found in the experimental (vegetarian) group compared to the control (conventional diet) group despite the similar advise on caloric restriction in both diets. The differences between the two groups will increase after an intensive physical exercise program.

DETAILED DESCRIPTION:
Open randomized study. Individuals with type 2 diabetes (n=60) will be recruited through newspaper advertisements and through advertisements in the hospital. They will be randomly assigned to a low-fat vegetarian diet or a diet following the guidelines of the Study Group on Diabetes and Nutrition of the European Association for the Study of Diabetes (DNSG) (21) with similar caloric restriction (-500 kcal/d). The participants will be followed for 12 weeks and then for another 12 weeks with the addition of intensive physical exercise. All meals during the 6 months will be provided.

ELIGIBILITY:
Inclusion Criteria:

1. Individuals with type 2 diabetes as defined by the criteria of the American Diabetes Association and recognized by WHO, Expert Committee on the Diagnosis and Classification of Diabetes Mellitus (19,20)
2. Concurrent T2 DM therapy: The use of oral hypoglycemic medication stable for the last 3 months
3. HbA1c ≥ 4 and ≤ 9.0 % (IFCC) ~ ≥ 6.0 and ≤ 11 % (DCCT)
4. Men and women who are 30 to 70 years of age
5. Body Mass Index (kg/m2) between 25 and 53
6. Informed Consent: a signed and dated written consent obtained from the subject before any procedures are performed
7. Willing to change dietary habits and to follow the prescribed diet and exercise program

Exclusion Criteria:

1. Current alcohol or drug abuse
2. Pregnancy, lactating
3. Unstable medical status
4. Diagnosis of Type 1 diabetes mellitus
5. Significant weight gain or loss (defined as ≥ 10% of total body weight) within the past 3 months prior to screening.
6. Pacemaker or metal in the body.

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2008-07; Primary Completion 2008-11 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
Insulin resistance | 6 months

SECONDARY OUTCOMES:
Visceral to subcutaneous fatty tissue ratio | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Terezie Pelikanova, MD, PhD, Principal Investigator — Head of the Diabetes Center
Locations (1):
- Institute for Clinical and Experimental Medicine, Prague, Czechia

REFERENCES:
- [Derived] Kahleova H, Tonstad S, Rosmus J, Fisar P, Mari A, Hill M, Pelikanova T. The effect of a vegetarian versus conventional hypocaloric diet on serum concentrations of persistent organic pollutants in patients with type 2 diabetes. Nutr Metab Cardiovasc Dis. 2016 May;26(5):430-8. doi: 10.1016/j.numecd.2016.01.008. Epub 2016 Jan 28. PMID 27107842
- [Derived] Kahleova H, Matoulek M, Malinska H, Oliyarnik O, Kazdova L, Neskudla T, Skoch A, Hajek M, Hill M, Kahle M, Pelikanova T. Vegetarian diet improves insulin resistance and oxidative stress markers more than conventional diet in subjects with Type 2 diabetes. Diabet Med. 2011 May;28(5):549-59. doi: 10.1111/j.1464-5491.2010.03209.x. PMID 21480966